CLINICAL TRIAL: NCT06319560
Title: Hydroxychloroquine as an Adjunct Therapy in the Management of Type 2 Diabetes in Pregnancy: A Randomised Controlled Trial
Brief Title: Hydroxychloroquine in Type 2 Diabetes During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2023-866
Record Dates: First submitted 2024-01-23; First posted 2024-03-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Diabetes in Pregnancy; Type 2 Diabetes
Keywords: diabetes; pregnancy; hydroxychloroquine
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine group (Experimental): Oral hydroxychloroquine 200mg daily will be prescribed to women in this group from recruitment (14-20 weeks) till delivery, in addition to their standard treatment
  Interventions: Drug: Hydroxychloroquine Oral Tablet
- Standard treatment group (No Intervention): Women will receive standard treatment for diabetes such as metformin and insulin.

INTERVENTIONS:
Drug: Hydroxychloroquine Oral Tablet — 200mg daily
  Other Names: plaquenil
  Arms: Hydroxychloroquine group

SUMMARY:
The goal of this clinical trial is to compare the use of hydroxychloroquine as an adjunct to the current treatment of pregnant women with Type 2 diabetes mellitus.

The main questions it aims to answer are:

* Does hydroxychloroquine improve the pregnancy outcomes in women with type 2 diabetes during pregnancy?
* Does hydroxychloroquine improve the inflammatory markers in women with type 2 diabetes during pregnancy? Participants will be randomised into the intervention and control group. The control group will be on standard treatment where as the intervention group will receive hydroxychloroquine as an adjunct of standard treatment

DETAILED DESCRIPTION:
This is a randomised clinical trial comparing 2 groups i.e type 2 diabetes complicating pregnancies on standard treatment alone which comprises of oral hypoglycaemic agent with or without insulin and those with added hydroxychloroquine 200mg daily. They will be recruited within 14-20 weeks gestation. Randomisation will be done using computer software program. At recruitment, blood is withdrawn to measure glycated haemoglobin (HbA1c), full blood count, fructosamine, Interleukin-6, Interleukin-10 and Tumour Necrosis Factor-alpha. These investigations will be repeated before delivery. Patients will monitor their blood glucose using staggered 7 points which consisting of pre-meals and 1 hour post-meals using their own glucometer. The optimum fasting level is 4-5.3 mmol/l, pre meal and pre bed levels of 4-6 mmol/l and 1 hour post meal level of 4-7.8 mmol/l. All participants are followed up every 2-4 weekly whereby home blood glucose monitoring will be reviewed. Fetal growth will be monitored via serial ultrasound and charted on the fetal growth chart. Patients' care will be done by the research team which consist of obstetrician, endocrinologist and diabetic educator. All patients will have eye assessment by the ophthalmologist prior to commencement of hydroxychloroquine.

All women will be delivered at 38 weeks or earlier if there are other concomitant problems such as fetal growth restriction or poorly controlled diabetes via induction of labour. The details of the delivery for both mother and neonates will be documented. At birth, the offsprings will be seen by the neonatologist who is also in the research team. After delivery, participants will be followed up in research clinic at 6 and 12 months together with the neonate. The height and weight of the infants will be measured in centimeter. Developmental milestones will be assessed according to the developmental milestones chart of Paediatric Protocols for Malaysian Hospitals 4th Edition 2019.

Compliance to hydroxychloroquine will be assessed at each follow up, whereby an indirect method of assessing adherence of participants in the hydroxychloroquine group will be made. Each participant will be asked whether they are still taking the study medication and are required to bring the remaining medication for tablet count. Participants with remaining of more than 20% of the scheduled medications will be considered as non-compliance and treated as drop-out. Participants will also be considered as drop-out when they are lost to follow-up, withdrawal of consent, non-compliance to hydroxychloroquine or a patient becomes ill due to drug adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Singleton
* Pregnant women with a confirmed diagnosis of type 2 Diabetes Mellitus

Exclusion Criteria:

* autoimmune disease such as Systemic Lupus Erythematosus or rheumatic disease
* chronic kidney disease
* fetal anomaly
* women on steroid therapy
* diabetic retinopathy
* known thalassaemia or thalassaemia carrier

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the serum glycated haemoglobin (HbA1c) between the two groups | From Day 1 up to 38 weeks of gestation
  Serum level of glycated haemoglobin (HbA1c) in percentage
To compare the serum fructosamine between the two groups | From Day 1 up to 38 weeks of gestation
  Serum level of fructosamine in nanogram per milliliter
To compare the serum interleukin-6 between the two groups | From Day 1 up to 38 weeks of gestation
  Serum level of interleukin-6 in nanogram per milliliter
To compare the serum interleukin-10 between the two groups | From Day 1 up to 38 weeks of gestation
  Serum level of interleukin-10 in nanogram per milliliter
To compare the serum tumour necrosis factor alpha between the two groups | From Day 1 up to 38 weeks of gestation
  Serum level of tumour necrosis factor alpha in nanogram per milliliter

SECONDARY OUTCOMES:
To compare the gestational age at delivery between the two groups | From recruitment up to 38 weeks of gestation
  Gestational age at delivery in weeks
Type of labour | From recruitment up to 38 weeks of gestation
  Onset of labour either spontaneous or induced
Mode of delivery | From recruitment up to 38 weeks of gestation
  Method of patient being delivered either vaginal or caesarean section
Postpartum haemorrhage | Immediately from delivery up to 42 days post delivery
  Total blood loss of more than 500 milliliters for vaginal delivery and 1000 milliliters for caesarean delivery
Obstetric anal sphincter injuries | Immediately from delivery up to 24 hours
  The number of patients who suffered third or fourth degree perineal tear
Neonatal birth weight at delivery | At delivery up to 24 hours
  Birth weight of the neonate in grams, Neonatal birth weight of more than 90th percentile based on Fenton birth weight chart will be considered as large for gestational age or more than 4000 grams will be considered as macrosomia
Shoulder dystocia | At delivery up to 24 hours
  Number of patient who experienced shoulder dystocia at delivery
Appearance, pulse, grimace, activity and respiration score of neonate at 5 minutes | At delivery up to 10 minutes after delivery
  Number of neonates with Apgar score of less than 7 at birth which is bad outcome
Number of neonates needing admission into neonatal intensive care unit | At delivery up to 7 days of life
  Admission of neonate into neonatal intensive care unit at birth
Height of the infant | At six and twelve months of age after delivery
  Height or length of the infant measured in centimetres
Weight of the infant | At six and twelve months of age after delivery
  Weight of the infant measured in grams
Hospital admission | From day 7 of life up to twelve months of age
  Numbers of infants required hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Rahana Abd Rahman, Principal Investigator — UKM
Locations (1):
- Antenatal clinic, UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basri NI, A Wahab N, Mohammed Nawi A, Ishak S, Murthi P, Abd Rahman R. Hydroxychloroquine as an adjunct therapy in the management of type 2 diabetes in pregnancy: study protocol for a randomised controlled trial. BMJ Open. 2026 Jan 20;16(1):e106653. doi: 10.1136/bmjopen-2025-106653. PMID 41558753